CLINICAL TRIAL: NCT00160251
Title: PEG-Intron/REBETOL vs PEG-Intron/ SCH 503034 With and Without Ribavirin in Chronic Hepatitis C Virus Genotype 1 (HCV-1) Peginterferon Alfa/Ribavirin Nonresponders: A SCH 503034 Dose-Finding Phase 2 Study
Brief Title: Boceprevir (SCH 503034) Plus Peg-Intron, With and Without Added Ribavirin, in Patients With Chronic Hepatitis C, Genotype 1, Who Did Not Respond to Previous Treatment With Peginterferon Alfa Plus Ribavirin (Study P03659AM2)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P03659
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2011-12-29 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Hepatitis C
Keywords: PEG-Intron; Ribavirin; Protease Inhibitor
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Arm 1A: PegIntron (PEG) + Ribavirin (RBV) (Active Comparator): A single dose of PEG is given first, followed 1 week later by PEG + RBV for 12 weeks. If HCV-RNA is undetected, PEG + RBV will continue for another 36 weeks.
  Interventions: Biological: PegIntron (PEG); Drug: Ribavirin (RBV)
- Arm 1B: PegIntron (PEG)+Ribavirin (RBV)+Boceprevir (BOC) 400 (Active Comparator): A single dose of PEG is given first, followed 1 week later by PEG + RBV for 12 weeks. If HCV-RNA is detectable, BOC 400 mg TID will be added for 36 weeks. By second protocol amendment to P03659, participants will be rolled over into Arm 8 for the remainder of the treatment period.
  Interventions: Drug: Boceprevir (BOC); Biological: PegIntron (PEG); Drug: Ribavirin (RBV)
- Arm 2: PegIntron (PEG) + Boceprevir (BOC) 100 (48 weeks) (Experimental): A single dose of PEG is given first, followed 1 week later by PEB + BOC 100 for 48 weeks. By second protocol amendment to P03659, participants will be rolled over into Arm 8 for the remainder of the treatment period.
  Interventions: Drug: Boceprevir (BOC); Biological: PegIntron (PEG)
- Arm 3: PegIntron (PEG) + Boceprevir (BOC) 200 (48 Weeks) (Experimental): A single dose of PEG is given first, followed 1 week later by PEG + BOC 200 for 48 weeks. By second protocol amendment to P03659, participants will be rolled over into Arm 8 for the remainder of the treatment period.
  Interventions: Drug: Boceprevir (BOC); Biological: PegIntron (PEG)
- Arm 4: PegIntron (PEG) + Boceprevir (BOC) 400 (48 weeks) (Experimental): A single dose of PEG is given first, followed 1 week later by PEG + BOC 400 for 48 weeks. By second protocol amendment to P03659, participants will be rolled over into Arm 8 for the remainder of the treatment period.
  Interventions: Drug: Boceprevir (BOC); Biological: PegIntron (PEG)
- Arm 5: PegIntron (PEG)+Ribavirin (RBV)+Boceprevir (BOC) 400 (Experimental): A single dose of PEG is given first, followed 1 week later by PEG + RBV + BOC 400 for 48 weeks. By second protocol amendment to P03659, participants will be rolled over into Arm 8 for the remainder of the treatment period.
  Interventions: Drug: Boceprevir (BOC); Biological: PegIntron (PEG); Drug: Ribavirin (RBV)
- Arm 6: PegIntron (PEG) + Boceprevir (BOC) 400 (24 Weeks) (Experimental): A single dose of PEG is given first, followed 1 week later by PEG + BOC 400 for 24 weeks. By second protocol amendment to P03659, participants will be rolled over into Arm 8 for the remainder of the treatment period.
  Interventions: Drug: Boceprevir (BOC); Biological: PegIntron (PEG)
- Arm 7: PegIntron (PEG) + Boceprevir (BOC) 800 (Experimental): By first protocol amendment to P03659, this non-randomized arm is added. A single dose of PEG is given first, followed 1 week later by PEG + BOC 800 for 24 weeks. By second protocol amendment to P03659, participants will be rolled over into Arm 8 for the remainder of the treatment period.
  Interventions: Drug: Boceprevir (BOC); Biological: PegIntron (PEG)
- Arm 8: PegIntron (PEG)+Ribavirin (RBV)+Boceprevir (BOC) 800 (Experimental): By second protocol amendment to P03659, participants from all arms except Arm 1A will be rolled over into PEG + RBV + BOC 800 for the remainder of the treatment period.
  Interventions: Drug: Boceprevir (BOC); Biological: PegIntron (PEG); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Boceprevir (BOC) — 100 or 200 mg capusles taken orally as 100 mg, 200 mg, 400 mg, or 800 mg TID
  Other Names: SCH 503034
  Arms: Arm 1B: PegIntron (PEG)+Ribavirin (RBV)+Boceprevir (BOC) 400; Arm 2: PegIntron (PEG) + Boceprevir (BOC) 100 (48 weeks); Arm 3: PegIntron (PEG) + Boceprevir (BOC) 200 (48 Weeks); Arm 4: PegIntron (PEG) + Boceprevir (BOC) 400 (48 weeks); Arm 5: PegIntron (PEG)+Ribavirin (RBV)+Boceprevir (BOC) 400; Arm 6: PegIntron (PEG) + Boceprevir (BOC) 400 (24 Weeks); Arm 7: PegIntron (PEG) + Boceprevir (BOC) 800; Arm 8: PegIntron (PEG)+Ribavirin (RBV)+Boceprevir (BOC) 800
Biological: PegIntron (PEG) — 1.5 mcg/kg weekly subcutaneously
Drug: Ribavirin (RBV) — 200 mg capsules taken twice daily (BID) (total daily dose of 800-1400 mg/day, depending on weight [weight-based dosing {WBD}])
  Arms: Arm 1A: PegIntron (PEG) + Ribavirin (RBV); Arm 1B: PegIntron (PEG)+Ribavirin (RBV)+Boceprevir (BOC) 400; Arm 5: PegIntron (PEG)+Ribavirin (RBV)+Boceprevir (BOC) 400; Arm 8: PegIntron (PEG)+Ribavirin (RBV)+Boceprevir (BOC) 800

SUMMARY:
The primary objective of this study is to determine the safe and effective dose range of boceprevir (SCH 503034) in combination with PEG-Intron in adult subjects who have chronic hepatitis C without cirrhosis, and who have failed an adequate course of combination therapy with peginterferon-alfa plus ribavirin. A secondary objective is to explore whether ribavirin provides an additional benefit when combined with PEG-Intron plus boceprevir.

ELIGIBILITY:
Key inclusion criteria:

* Documented infection with chronic hepatitis C (CHC), genotype 1.
* Documented failure to respond to an adequate course of treatment (minimum 12 weeks) with peginterferon-alfa plus ribavirin (failure defined as <2 log drop in HCV-RNA after 12 weeks of therapy or those who never become Hepatitis C Virus Ribonucleic Acid (HCV)-RNA negative)
* No evidence of cirrhosis on liver biopsy.
* Results of physical examination and laboratory tests within specified ranges.
* Abstinence from use of abused substances.

Key exclusion criteria:

* Women who are pregnant or nursing a child.
* Patients with cirrhosis, co-infection with Hepatitis B or human immunodeficiency virus (HIV), and African-American patients (by protocol amendment 2, African-American patients can enroll).
* Previous treatment with any Hepatitis C Virus (HCV) polymerase or protease inhibitor.
* Patients who relapsed following response to previous treatment.
* Evidence of advanced liver disease, or liver disease from a cause other than CHC.
* Pre-existing psychiatric condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1A: PEG + RBV; Arm 5: PEG + RBV + BOC 400; ARM 4+6: PEG + BOC 400 (24 + 48 Weeks): A single dose of PEG was given first, followed 1 week A single dose of PEG was given first, followed 1 week later by PEG + RBV + BOC 400. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- Arm 1B: PEG + RBV + BOC: A single dose of PEG was given first, followed 1 week later by PEG + RBV for 12 weeks. If HCV-RNA was detectable, BOC 400 was added for another 36 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- Arm 2: PEG + BOC 100 (48 Weeks): A single dose of PEG was given first, followed 1 week later by PEG + BOC 100 for 48 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- Arm 3: PEG + BOC 200 (48 Weeks): A single dose of PEG was given first, followed 1 week later by PEG + BOC 200 for 48 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- Arm 7: PEG + BOC 800: A single dose of PEG was given first, followed 1 week later by PEG + BOC 800. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- Arm 8: PEG + RBV + BOC 800: By protocol amendment 2, participants from all arms except Arm 1A were rolled over into PEG + RBV + BOC 800 for the remainder of the treatment period.
Period: Prior to Amendment 2
Arm/Group | Arm 1A: PEG + RBV | Arm 1B: PEG + RBV + BOC | Arm 2: PEG + BOC 100 (48 Weeks) | Arm 3: PEG + BOC 200 (48 Weeks) | Arm 5: PEG + RBV + BOC 400 | ARM 4+6: PEG + BOC 400 (24 + 48 Weeks) | Arm 7: PEG + BOC 800 | Arm 8: PEG + RBV + BOC 800
Started | 15 | 34 | 48 | 49 | 49 | 97 | 65 | 0
Completed | 6 | 28 | 4 | 9 | 21 | 14 | 61 | 0
Not Completed | 9 | 6 | 44 | 40 | 28 | 83 | 4 | 0
Not completed — Adverse Event | 2 | 1 | 3 | 1 | 1 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 4 | 37 | 35 | 24 | 55 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 3 | 4 | 2 | 3 | 3 | 0
Not completed — Noncompliance with protocol | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Completed Treatment Phase | 3 | 0 | 0 | 0 | 0 | 23 | 0 | 0
Period: Post-amendment 2
Arm/Group | Arm 1A: PEG + RBV | Arm 1B: PEG + RBV + BOC | Arm 2: PEG + BOC 100 (48 Weeks) | Arm 3: PEG + BOC 200 (48 Weeks) | Arm 5: PEG + RBV + BOC 400 | ARM 4+6: PEG + BOC 400 (24 + 48 Weeks) | Arm 7: PEG + BOC 800 | Arm 8: PEG + RBV + BOC 800
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 143
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 88
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 55
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24
Not completed — Lost to follow-up/withdrawal by subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Arm 1A: PEG + RBV OR Arm 1B: PEG + RBV + BOC 400: Arm 1A: A single dose of PEG was given first, followed 1 week later by PEG + RBV for 12 weeks. If participant was HCV-RNA negative, PEG + RBV was continued for another 36 weeks.
  Arm 1B: A single dose of PEG was given first, followed 1 week later by PEG + RBV for 12 weeks. If HCV-RNA was detectable, BOC 400 was added for another 36 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- Arm 5: PEG + RBV + BOC 400: A single dose of PEG was given first, followed 1 week later by PEG + RBV + BOC 400. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- Arms 4 + 6: PEG + BOC 400 (24 + 48 Weeks): A single dose of PEG was given first, followed 1 week later by PEG + BOC (24 or 48 weeks). By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- Total: Total of all reporting groups
Arm/Group | Arm 1A: PEG + RBV OR Arm 1B: PEG + RBV + BOC 400 | Arm 2: PEG + BOC 100 (48 Weeks) | Arm 3: PEG + BOC 200 (48 Weeks) | Arm 5: PEG + RBV + BOC 400 | Arms 4 + 6: PEG + BOC 400 (24 + 48 Weeks) | Arm 7: PEG + BOC 800 | Total
Number analyzed (Participants) | 49 | 48 | 49 | 49 | 97 | 65 | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (9.7) | 51.6 (7.0) | 48.6 (9.4) | 48.2 (8.9) | 49.2 (8.7) | 50.4 (7.3) | 49.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 14 | 21 | 37 | 24 | 134
  Male | 32 | 27 | 35 | 28 | 60 | 41 | 223

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Were Hepatitis C Virus Ribonucleic Acid (HCV-RNA) Negative at the End of Treatment (EoT)
Description: Sustained Viral Response (SVR) was defined as the percentage of participants with HCV-RNA undetectable at the follow-up Week 24.
  All percentages were based on the total number of participants originally randomized/enrolled to that particular arm.
  For Arm 1B, the denominator for the percentages was the number who received at least 1 dose of BOC.
  Arm 1A was not analyzed.
Time Frame: Baseline up to Week 49
Population: For PEG + RBV + BOC number of participants was number who received at least one dose of BOC. For all others, it was number of randomized participants. The PEG + BOC 800 arm was not randomized.
Measure: Number; unit: Percent of participants
Groups:
- Arm 1B: PEG + RBV + BOC 400: A single dose of PEG was given first, followed 1 week later by PEG + RBV for 12 weeks. If HCV-RNA was detectable, BOC 400 was added for another 36 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
Arm/Group | Arm 1B: PEG + RBV + BOC 400 | Arm 2: PEG + BOC 100 (48 Weeks) | Arm 3: PEG + BOC 200 (48 Weeks) | Arms 4 + 6: PEG + BOC 400 (24 + 48 Weeks) | Arm 5: PEG + RBV + BOC 400 | Arm 7: PEG + BOC 800
Number analyzed (Participants) | 40 | 48 | 49 | 97 | 49 | 65
Percent of participants | 35.0 | 6.3 | 16.3 | 13.4 | 20.4 | 21.5

2. Secondary Outcome: Percent of Participants Who Achieved Sustained Viral Response (SVR) by Time to First Negative HCV-RNA
Description: Percentage of participants who became HCV-RNA undetectable within the first 13 weeks and subsequently became HCV-RNA positive were not considered negative for this analysis.
Time Frame: Baseline up to Week 73 [24 weeks after EoT]
Population: Number of participants across all treatment arms who achieved negative HCV-RNA
Measure: Number; unit: Percent of participants
Groups:
- 0 to ≤ 4 Weeks to First Negative HCV-RNA Group: Participants who achieved first negative HCV RNA within the first 4 weeks of treatment.
- >4 to 8 Weeks to First Negative HCV-RNA Group: Participants who achieved first negative HCV RNA between weeks 4 to 8.
- >8 to 12 Weeks to First Negative HCV-RNA Group: Participants who achieved first negative HCV RNA between weeks 8 to 12.
- >12 to 36 Weeks to First Negative HCV-RNA Group: Participants who achieved first negative HCV RNA between weeks 12 to 36.
Arm/Group | 0 to ≤ 4 Weeks to First Negative HCV-RNA Group | >4 to 8 Weeks to First Negative HCV-RNA Group | >8 to 12 Weeks to First Negative HCV-RNA Group | >12 to 36 Weeks to First Negative HCV-RNA Group
Number analyzed (Participants) | 33 | 12 | 6 | 11
Percent of participants | 58 | 33 | 33 | 0

3. Secondary Outcome: Percentage of Participants Who Were HCV-RNA Negative at EoT After Receiving 1 Week of Treatment With PegIntron (PEG) by Log Drop
Description: For each log drop category (<0, 0 to 0.5, 0.5 to <1, 1 to <1.5, ≥1.5, and Missing), the percentage of participants receiving combination therapy who were HCV-RNA negative at EoT (Week 49) was calculated as follows:
  Number of participants in a log category who were HCV-RNA negative divided by the total number of participants in that log drop category (n).
  Percentages were NOT derived using treatment arm N values. The sum of the n values for all 6 log drop categories within a treatment arm equals the overall N for that treatment group.
Time Frame: Week 1 and Week 49
Population: N=Number of Participants Analyzed, n=number of participants in each log category group. The PEG + BOC 100, 200, or 400 arm combined the following treatment arms: Arm 2 PEG + BOC 100 (48 weeks), Arm 3 PEG + BOC 200 (48 weeks), Arm 4 PEG + BOC 400 (48 weeks), Arm 6 PEG + BOC 400 (24 weeks).
Measure: Number; unit: Percent of participants
Groups:
- Arms 2, 3, 4, 6: PEG + BOC 100, 200, or 400: A single dose of PEG was given first, followed 1 week later by PEG + BOC. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
Arm/Group | Arms 2, 3, 4, 6: PEG + BOC 100, 200, or 400 | Arm 5: PEG + RBV + BOC 400 | Arm 7: PEG + BOC 800
Number analyzed (Participants) | 194 | 49 | 65
Percent of participants
  Log drop <0 (Arm2-4,6 n=21/Arm5 n=6/Arm7 n=3) | 9.5 | 16.7 | 1
  Log drop 0-0.5 (Arm2-4,6 n=55/Arm5 n=17/Arm7 n=16) | 1.8 | 17.6 | 18.8
  Log drop 0.5to<1(Arm2-4,6 n=73/Arm5 n=11/Arm7 n=9) | 12.3 | 9.1 | 0
  Log drop 1to<1.5(Arm2-4,6 n=31/Arm5 n=9/Arm7 n=18) | 25.8 | 33.3 | 16.7
  Log drop ≥1.5 (Arm2-4,6 n=12/Arm5 n=4/Arm7 n=18) | 33.3 | 50.0 | 44.4
  Missing (Arm2-4,6 n=2/Arm5 n=2/Arm7 n=1) | 0 | 0 | 0

4. Secondary Outcome: Percent of Participants With Virologic Response Prior to Amendment 2
Description: Virologic response was defined as the percentage of participants with Hepatitis C Virus Ribonucleic Acid (HCV-RNA) ≤10,000 IU/mL.
Time Frame: Week 3, Week 5, Week 13
Measure: Number; unit: Percent of participants
Groups:
- Arm 1A: PEG + RBV and Arm 1B: PEG + RBV + BOC 400: Arm 1A: A single dose of PEG was given first, followed 1 week later by PEG + RBV for 12 weeks. If participant was HCV-RNA negative, PEG + RBV was continued for another 36 weeks.
  Arm 1B: A single dose of PEG was given first, followed 1 week later by PEG + RBV for 12 weeks. If HCV-RNA was detectable, BOC 400 was added for another 36 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
Arm/Group | Arm 1A: PEG + RBV and Arm 1B: PEG + RBV + BOC 400 | Arm 2: PEG + BOC 100 (48 Weeks) | Arm 3: PEG + BOC 200 (48 Weeks) | Arm 5: PEG + RBV + BOC 400 | Arms 4 + 6: PEG + BOC 400 (24 + 48 Weeks) | Arm 7: PEG + BOC 800
Number analyzed (Participants) | 49 | 48 | 49 | 49 | 97 | 65
Percent of participants
  Week 3 | 4.1 | 0.0 | 0.0 | 0 | 5.2 | 4.6
  Week 5 | 4.1 | 0.0 | 8.2 | 12.2 | 9.3 | 15.4
  Week 13 | 6.1 | 2.1 | 14.3 | 30.6 | 13.4 | 0

5. Secondary Outcome: Peak Plasma Concentration of Boceprevir (BOC)
Description: All plasma samples were assayed using a validated liquid chromatography with tandem mass spectrometric detection (LCMS/MS) method.
Time Frame: All visits during treatment (baseline to Week 49) except Day 1 of Week 1
Population: Participants were only included in the analysis if the recorded previous dose of boceprevir was taken < 8.5 hours prior to sample collection. Participants also must have started BOC treatment or amendment 2 dosing more than 1 week prior to sample collection.
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- BOC 100 mg Dose: A single dose of PEG was given first, followed 1 week later by Arm 2 (PEG + BOC 100). By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- BOC 200 mg Dose: A single dose of PEG was given first, followed 1 week later by Arm 3 (PEG + BOC 200). By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- BOC 400 mg Dose: A single dose of PEG was given first, followed 1 week later by Arms 1B, 4, 5, 6, or 7. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- BOC 800 mg Dose: A single dose of PEG was given first, followed 1 week later by PEG + BOC 800 or PEG + RBV + BOC 800. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
Arm/Group | BOC 100 mg Dose | BOC 200 mg Dose | BOC 400 mg Dose | BOC 800 mg Dose
Number analyzed (Participants) | 29 | 24 | 62 | 64
ng/mL | 203 (5) | 427 (18) | 704 (16) | 1312 (45)

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve of Boceprevir Plasma Concentration for an 8-hour Dosing Period
Description: All plasma samples were assayed using a validated liquid chromatography with tandem mass spectrometric detection (LCMS/MS) method.
  The dosing interval of 8 hours is represented as the hr in the unit of measure.
Time Frame: All visits during treatment (baseline to Week 49) except Day 1 of Week 1
Population: as for outcome 5
Measure: Mean (Standard Error); unit: ng*hr/mL
Arm/Group | BOC 100 mg Dose | BOC 200 mg Dose | BOC 400 mg Dose | BOC 800 mg Dose
Number analyzed (Participants) | 29 | 24 | 62 | 64
ng*hr/mL | 1042 (25) | 2184 (181) | 3633 (88) | 6276 (337)

7. Secondary Outcome: Trough Plasma Concentration Level
Description: as for outcome 5
Time Frame: All visits during treatment (baseline to Week 49) except Day 1 of Week 1
Population: as for outcome 5
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | BOC 100 mg Dose | BOC 200 mg Dose | BOC 400 mg Dose | BOC 800 mg Dose
Number analyzed (Participants) | 29 | 24 | 62 | 64
ng/mL | 56.7 (3) | 133.0 (27) | 214.0 (10) | 355 (42)

8. Secondary Outcome: Change in Alanine Aminotransferase (ALT) Levels
Description: Change in ALT levels during initial treatment regimen and after rolling into amendment 2 as compared to baseline.
Time Frame: Baseline up to dosing change (> 25 weeks)
Population: Only participants with at least one value for the laboratory test were included.
Measure: Number; unit: Participants
Groups:
- Arm 1A: PEG + RBV: Arm 1A: A single dose of PEG was given first, followed 1 week later by PEG + RBV for 12 weeks. If participant was HCV-RNA negative, PEG + RBV was continued for another 36 weeks.
- Arm 1B: PEG + RBV + BOC 400: Arm 1B: A single dose of PEG was given first, followed 1 week later by PEG + RBV for 12 weeks. If HCV-RNA was detectable, BOC 400 was added for another 36 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- Arm 3: PEG + BOC 200: A single dose of PEG was given first, followed 1 week later by PEG + BOC 200 for 48 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
Arm/Group | Arm 1A: PEG + RBV | Arm 1B: PEG + RBV + BOC 400 | Arm 2: PEG + BOC 100 (48 Weeks) | Arm 3: PEG + BOC 200 | Arm 5: PEG + RBV + BOC 400 | Arms 4 + 6: PEG + BOC 400 (24 + 48 Weeks) | Arm 7: PEG + BOC 800 | Arm 8: PEG + RBV + BOC 800
Number analyzed (Participants) | 15 | 34 | 48 | 47 | 48 | 97 | 64 | 143
Participants
  <2.00 x baseline ALT value | 14 | 33 | 45 | 43 | 47 | 84 | 61 | 119
  2.00-2.09 x baseline ALT value | 1 | 1 | 1 | 1 | 0 | 4 | 0 | 4
  2.10-5.09 x baseline ALT value | 0 | 0 | 2 | 3 | 1 | 9 | 3 | 18
  5.10-10.0 x baseline ALT value | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  >10.0 x baseline ALT value | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

9. Secondary Outcome: Number of Participants Who Were HCV-RNA Negative During Amendment 2 (AM2) for Those Who Started on Arms 2 (PEG+BOC 100), 3 (PEG+BOC 200), 4 (PEG+BOC 400 [48 Weeks]), 6 (PEG+BOC 400 [24 Weeks])
Description: Log drop at baseline of dosing change = difference of log viral loads between baseline (closest to the treatment begin date) and dosing change baseline (virology value closest to the dosing change begin date).
Time Frame: From dosing change to end of follow-up (Week 73)(up to 48 weeks)
Population: All participants, per the second amendment to P03659, with significant HCV-RNA decrease (HCV_RNA ≤ 10,000 IU) switched to continuing triple therapy.
Measure: Number; unit: Participants
Groups:
- Log Drop 0 to <1; Log Drop 1 to <2; Log Drop 2 to <3; Log Drop 3 to <4; Log Drop 4 to <5; Log Drop ≥5: All arms were given single dose of PEG first, followed 1 week later by PEG + BOC 100 for 48 weeks for Arm 2 (PEG+BOC 100), followed by PEG + BOC 200 for 48 weeks for Arm 3 (PEG+BOC 200), followed by PEG + BOC (24 or 48 weeks) for Arm 4 (PEG+BOC 400 [48 weeks]) and Arm 6 (PEG+BOC 400 [24 weeks]). By protocol amendment 2, participants were switched to an increased dose of BOC 800 TID plus RBV with PEG for an additional 24 Weeks of Treatment.
Arm/Group | Log Drop 0 to <1 | Log Drop 1 to <2 | Log Drop 2 to <3 | Log Drop 3 to <4 | Log Drop 4 to <5 | Log Drop ≥5
Number analyzed (Participants) | 4 | 2 | 2 | 4 | 12 | 3
Participants
  Week 3 after dosing change | 0 | 0 | 0 | 4 | 11 | 2
  Week 6 after dosing change | 0 | 0 | 0 | 4 | 11 | 1
  Week 9 after dosing change | 0 | 0 | 0 | 4 | 9 | 1
  Week 12 after dosing change | 0 | 0 | 0 | 4 | 9 | 1
  Week 18 after dosing change | 1 | 0 | 1 | 4 | 11 | 1
  Week 24 after dosing change | 1 | 0 | 1 | 4 | 12 | 1
  End of treatment | 1 | 0 | 1 | 4 | 11 | 1
  Follow-up Week 4 after dosing change | 0 | 0 | 0 | 4 | 8 | 1
  Follow-up Week 8 after dosing change | 0 | 0 | 0 | 4 | 6 | 1
  Follow-up Week 12 after dosing change | 0 | 0 | 0 | 4 | 6 | 1
  Follow-up Week 24 after dosing change | 0 | 0 | 0 | 4 | 7 | 1
  End of follow-up after dosing change | 0 | 0 | 0 | 4 | 7 | 1

10. Secondary Outcome: Number of Participants Who Were HCV-RNA Negative During Amendment 2 (AM2) for Those Who Started on PegIntron (PEG) + Rebetol (RVB) + Boceprevir (BOC) 400 (Arm 5)
Description: as for outcome 9
Time Frame: From dosing change to end of follow-up (Week 73)(up to 48 weeks)
Population: as for outcome 9
Measure: Number; unit: Participants
Groups:
- Log Drop 1 to <2; Log Drop 2 to <3; Log Drop 3 to <4; Log Drop 4 to <5; Log Drop ≥5: Arm 5: A single dose of PEG first, followed 1 week later by PEG + RBV + BOC 400 for 48 weeks. By protocol amendment 2, participants were switched to an increased dose of BOC 800 plus RBV with PEG for an additional 24 Weeks of Treatment.
Arm/Group | Log Drop 1 to <2 | Log Drop 2 to <3 | Log Drop 3 to <4 | Log Drop 4 to <5 | Log Drop ≥5
Number analyzed (Participants) | 1 | 1 | 4 | 14 | 1
Participants
  Week 3 after dosing change | 0 | 0 | 3 | 12 | 1
  Week 6 after dosing change | 0 | 0 | 3 | 10 | 0
  Week 9 after dosing change | 0 | 0 | 3 | 10 | 0
  Week 12 after dosing change | 0 | 0 | 3 | 9 | 0
  Week 18 after dosing change | 0 | 0 | 2 | 6 | 0
  Week 24 after dosing change | 0 | 0 | 3 | 5 | 0
  End of treatment | 0 | 0 | 3 | 7 | 0
  Follow-up Week 4 after dosing change | 0 | 0 | 3 | 6 | 0
  Follow-up Week 8 after dosing change | 0 | 0 | 3 | 4 | 0
  Follow-up Week 12 after dosing change | 0 | 0 | 2 | 5 | 0
  Follow-up Week 24 after dosing change | 0 | 0 | 3 | 4 | 0
  End of follow-up after dosing change | 0 | 0 | 3 | 4 | 0

11. Secondary Outcome: Number of Participants Who Were HCV-RNA Negative During Amendment 2 (AM2) for Those Who Started on PegIntron (PEG) + Boceprevir (BOC) 800 (Arm 7)
Description: as for outcome 9
Time Frame: From dosing change to end of follow-up (Week 73) (up to 48 weeks)
Population: as for outcome 9
Measure: Number; unit: Participants
Groups:
- Log Drop <0; Log Drop 0 to <1; Log Drop 1 to <2; Log Drop 2 to <3; Log Drop 3 to <4; Log Drop 4 to <5; Log Drop ≥5; Missing Data: Arm 7: A single dose of PEG was given first, followed 1 week later by PEG + BOC 800. By protocol amendment 2, participants were switched to PEG + RBV + BOC 800 for an additional 24 Weeks of Treatment.
Arm/Group | Log Drop <0 | Log Drop 0 to <1 | Log Drop 1 to <2 | Log Drop 2 to <3 | Log Drop 3 to <4 | Log Drop 4 to <5 | Log Drop ≥5 | Missing Data
Number analyzed (Participants) | 2 | 12 | 12 | 5 | 10 | 9 | 6 | 5
Participants
  Week 3 after dosing change | 0 | 0 | 0 | 0 | 5 | 7 | 4 | 3
  Week 6 after dosing change | 0 | 0 | 0 | 0 | 3 | 5 | 4 | 1
  Week 9 after dosing change | 0 | 0 | 0 | 0 | 5 | 7 | 3 | 1
  Week 12 after dosing change | 0 | 0 | 0 | 1 | 4 | 5 | 4 | 2
  Week 18 after dosing change | 0 | 0 | 0 | 1 | 5 | 3 | 4 | 2
  Week 24 after dosing change | 0 | 0 | 1 | 1 | 4 | 3 | 4 | 1
  End of treatment | 0 | 0 | 1 | 1 | 4 | 3 | 4 | 1
  Follow-up Week 4 after dosing change | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
  Follow-up Week 8 after dosing change | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Follow-up Week 12 after dosing change | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Follow-up Week 24 after dosing change | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  End of follow-up after dosing change | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0

12. Primary Outcome: Percent of Participants Who Achieved Sustained Virologic Response (SVR)
Description: SVR was defined as the percentage of participants with Hepatitis C Virus Ribonucleic Acid (HCV-RNA) undetectable at the follow-up Week 24.
  All percentages were based on the total number of participants originally randomized/enrolled to that particular arm.
  For Arm 1B, the denominator for the percentages was the number who received at least 1 dose of BOC.
  Arm 1A was not analyzed.
Time Frame: Baseline up to Week 73 [24 weeks after end of treatment (EoT)]
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Arm 1B: PEG + RBV + BOC 400 | Arm 2: PEG + BOC 100 (48 Weeks) | Arm 3: PEG + BOC 200 (48 Weeks) | Arms 4 + 6: PEG + BOC 400 (24 + 48 Weeks) | Arm 5: PEG + RBV + BOC 400 | Arm 7: PEG + BOC 800
Number analyzed (Participants) | 40 | 48 | 49 | 97 | 49 | 65
Percent of participants | 7.5 | 2.1 | 12.2 | 5.2 | 14.3 | 4.6

ADVERSE EVENTS:
Groups:
- PEG + RBV: Arm 1A: A single dose of PEG was given first, followed 1 week later by PEG + RBV for 12 weeks. If participant was HCV-RNA negative, PEG + RBV was continued for another 36 weeks.
- PEG + RBV + BOC 400 (24 Weeks): Arm 1B: A single dose of PEG was given first, followed 1 week later by PEG + RBV for 12 weeks. If HCV-RNA was detectable, BOC 400 was added for another 36 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- PEG + BOC 100 (48 Weeks): Arm 2: A single dose of PEG was given first, followed 1 week later by PEG + BOC 100 for 48 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- PEG + BOC 200 (48 Weeks): Arm 3: A single dose of PEG was given first, followed 1 week later by PEG + BOC 200 for 48 weeks. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- PEG + RBV + BOC 400 (48 Weeks): Arm 5: A single dose of PEG was given first, followed 1 week later by PEG + RBV + BOC 400. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- PEG + BOC 400 (24 + 48 Weeks): Arms 4 + 6: A single dose of PEG was given first, followed 1 week later by PEG + BOC (24 or 48 weeks). By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- PEG + BOC 800 (24 Weeks): Arm 7: A single dose of PEG was given first, followed 1 week later by PEG + BOC 800. By protocol amendment 2, participants were rolled over into Arm 8 for the remainder of the treatment period.
- PEG + RBV + BOC 800: Arm 8: By protocol amendment 2, participants from all arms except Arm 1A were rolled over into PEG + RBV + BOC 800 for the remainder of the treatment period.
Arm/Group | PEG + RBV | PEG + RBV + BOC 400 (24 Weeks) | PEG + BOC 100 (48 Weeks) | PEG + BOC 200 (48 Weeks) | PEG + RBV + BOC 400 (48 Weeks) | PEG + BOC 400 (24 + 48 Weeks) | PEG + BOC 800 (24 Weeks) | PEG + RBV + BOC 800
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/34 | 2/48 | 4/49 | 2/49 | 4/97 | 3/65 | 12/143
Other Adverse Events (participants affected / at risk) | 14/15 | 33/34 | 48/48 | 48/49 | 47/49 | 96/97 | 64/65 | 136/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG + RBV (N=15) | PEG + RBV + BOC 400 (24 Weeks) (N=34) | PEG + BOC 100 (48 Weeks) (N=48) | PEG + BOC 200 (48 Weeks) (N=49) | PEG + RBV + BOC 400 (48 Weeks) (N=49) | PEG + BOC 400 (24 + 48 Weeks) (N=97) | PEG + BOC 800 (24 Weeks) (N=65) | PEG + RBV + BOC 800 (N=143)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALCOHOLIC PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHRONIC HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MASTOIDITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FOOD INTOLERANCE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADIAL NERVE PALSY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROSTATITIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIVER TRANSPLANT (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG + RBV (N=15) | PEG + RBV + BOC 400 (24 Weeks) (N=34) | PEG + BOC 100 (48 Weeks) (N=48) | PEG + BOC 200 (48 Weeks) (N=49) | PEG + RBV + BOC 400 (48 Weeks) (N=49) | PEG + BOC 400 (24 + 48 Weeks) (N=97) | PEG + BOC 800 (24 Weeks) (N=65) | PEG + RBV + BOC 800 (N=143)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 8 (12) | 1 (1) | 2 (2) | 54 (58)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 2 (6) | 0 (0) | 7 (13)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (4) | 3 (3) | 5 (7) | 5 (5) | 9 (16) | 12 (20) | 9 (10) | 25 (37)
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 2 (3)
PALPITATIONS (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (6)
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 6 (8)
DRY EYE (Eye disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
EYE IRRITATION (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
EYE PRURITUS (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 3 (3)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (5) | 2 (3) | 4 (4) | 5 (6) | 3 (3) | 4 (4)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 4 (4) | 9 (12) | 9 (13) | 5 (6) | 17 (21) | 1 (1) | 11 (14)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 8 (10)
DIARRHOEA (Gastrointestinal disorders) | 6 (9) | 7 (8) | 11 (14) | 11 (13) | 10 (16) | 29 (41) | 21 (23) | 13 (14)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 3 (3) | 7 (8) | 3 (3) | 5 (5)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 2 (3) | 5 (5) | 2 (2) | 5 (5) | 6 (6) | 2 (2) | 4 (6)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 6 (6) | 0 (0) | 1 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 5 (5)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 6 (7) | 9 (12) | 15 (17) | 13 (14) | 22 (31) | 32 (41) | 23 (23) | 22 (30)
ORAL MUCOSAL BLISTERING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
VOMITING (Gastrointestinal disorders) | 2 (3) | 4 (4) | 7 (10) | 5 (5) | 10 (15) | 11 (12) | 6 (6) | 9 (14)
ASTHENIA (General disorders) | 1 (1) | 9 (9) | 8 (9) | 7 (12) | 10 (15) | 20 (31) | 4 (4) | 7 (7)
CHEST PAIN (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
CHILLS (General disorders) | 4 (5) | 11 (16) | 19 (20) | 20 (22) | 19 (24) | 28 (33) | 27 (33) | 3 (3)
FATIGUE (General disorders) | 10 (12) | 14 (16) | 25 (31) | 31 (39) | 24 (33) | 45 (58) | 40 (48) | 38 (43)
FEELING HOT (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 5 (5) | 6 (6) | 7 (8) | 12 (13) | 10 (13) | 21 (24) | 15 (15) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 4 (4) | 4 (4) | 10 (11) | 10 (10) | 11 (11) | 15 (17) | 10 (10) | 1 (1)
INJECTION SITE RASH (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INJECTION SITE REACTION (General disorders) | 2 (2) | 6 (6) | 9 (9) | 5 (5) | 5 (5) | 9 (9) | 7 (7) | 0 (0)
IRRITABILITY (General disorders) | 3 (3) | 9 (9) | 7 (7) | 4 (8) | 9 (10) | 12 (14) | 7 (8) | 7 (7)
MALAISE (General disorders) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
PAIN (General disorders) | 1 (1) | 4 (6) | 4 (5) | 3 (3) | 3 (4) | 8 (8) | 3 (3) | 1 (1)
PYREXIA (General disorders) | 4 (4) | 13 (15) | 19 (26) | 17 (22) | 20 (26) | 30 (39) | 23 (27) | 6 (6)
HEPATOMEGALY (Hepatobiliary disorders) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 5 (5) | 9 (10) | 4 (4) | 1 (1)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
BRONCHITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 5 (5)
FOLLICULITIS (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 4 (4) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (2) | 4 (6) | 0 (0) | 2 (2)
ORAL HERPES (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 1 (2) | 1 (1) | 7 (7) | 1 (1) | 3 (3)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (3) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 6 (7) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 2 (5)
VIRAL PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 5 (5)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
SUNBURN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 9 (10)
WEIGHT DECREASED (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 6 (7)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 6 (6) | 6 (7) | 3 (3) | 4 (4) | 4 (4) | 5 (5)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 4 (5) | 5 (5) | 6 (6) | 8 (8)
HYPERINSULINISM (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (10) | 17 (28) | 15 (24) | 17 (18) | 35 (46) | 15 (22) | 8 (8)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 4 (4) | 6 (6) | 5 (5) | 21 (21) | 10 (10) | 9 (9)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (5) | 1 (2) | 3 (3) | 3 (3) | 1 (2) | 6 (6)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (10) | 23 (28) | 16 (20) | 16 (20) | 37 (39) | 26 (32) | 6 (7)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 5 (6) | 1 (1) | 5 (6)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 0 (0) | 5 (6) | 5 (5) | 2 (2) | 4 (5) | 4 (4) | 5 (5)
DIZZINESS (Nervous system disorders) | 2 (2) | 10 (10) | 10 (13) | 5 (5) | 4 (4) | 7 (9) | 6 (7) | 18 (23)
DYSGEUSIA (Nervous system disorders) | 3 (3) | 4 (4) | 3 (4) | 2 (2) | 13 (16) | 23 (26) | 31 (33) | 14 (14)
HEADACHE (Nervous system disorders) | 7 (9) | 20 (24) | 30 (39) | 28 (47) | 25 (37) | 52 (65) | 33 (43) | 11 (16)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 2 (2) | 3 (3)
HYPOKINESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 2 (2) | 0 (0)
SPEECH DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 3 (4) | 2 (2) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (3) | 4 (4) | 6 (7) | 4 (4) | 5 (5) | 8 (10) | 2 (2) | 6 (6)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
DEPRESSION (Psychiatric disorders) | 4 (5) | 4 (5) | 12 (13) | 8 (9) | 16 (16) | 18 (19) | 5 (7) | 22 (26)
INITIAL INSOMNIA (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 4 (4) | 9 (12) | 12 (14) | 11 (13) | 15 (18) | 20 (23) | 10 (10) | 23 (23)
MOOD SWINGS (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NERVOUSNESS (Psychiatric disorders) | 1 (1) | 3 (3) | 2 (4) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
SLEEP DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
SEXUAL DYSFUNCTION (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (12) | 9 (9) | 5 (5) | 7 (8) | 10 (12) | 6 (7) | 17 (20)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 6 (9) | 6 (6) | 11 (14) | 11 (11) | 0 (0) | 19 (21)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 11 (11)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 2 (3) | 3 (3) | 2 (2) | 3 (4) | 2 (12) | 0 (0) | 3 (26)
INCREASED UPPER AIRWAY SECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 2 (3)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 5 (6) | 2 (3) | 5 (6) | 7 (7) | 3 (3) | 7 (7)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6) | 10 (10) | 4 (5) | 17 (18) | 21 (21) | 2 (2) | 19 (19)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (9) | 6 (7) | 5 (5) | 8 (8) | 10 (10) | 2 (2) | 3 (4)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 2 (3) | 3 (3) | 3 (3) | 4 (5) | 4 (4) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
PALMAR ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (12) | 8 (10) | 4 (4) | 5 (5) | 9 (9) | 2 (2) | 15 (15)
RASH (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4) | 5 (5) | 3 (3) | 8 (12) | 9 (10) | 2 (2) | 9 (10)
SPIDER NAEVUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CYST DRAINAGE (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 2 (3) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The implementation of amendment 2 led to changes in boceprevir dose in all treatment arms and different overall lengths of therapy within the same treatment arm, making the SVR endpoint uninterpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator (PI) agrees to provide review copies to the sponsor 30 days prior to submission. The sponsor shall have editorial rights and the right to review and comment on the data analysis and presentation with regard to proprietary information, accuracy of information, and to ensure that the presentation is fairly balanced and in compliance with regulations. If the parties disagree, the PI agrees to meet with the sponsor to discuss and resolve any such issues or disagreement.